CLINICAL TRIAL: NCT06921408
Title: Retrospective Identification of Scintigraphic Cardiac Amyloidosis Using Deep Learning-based Model
Brief Title: Retrospective Identification of Scintigraphic Cardiac Amyloidosis (RISCA)
Acronym: RISCA
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Lille (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 2024_0111; ID RCB Number (Other: 2024-A01194-43)
Record Dates: First submitted 2025-04-03; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Cardiac Amyloidosis; Transthyretin Amyloidosis
Keywords: Cardiac Amyloidosis; Bone Scintigraphy; Deep learning
MeSH Terms: conditions — Amyloid Neuropathies, Familial; Amyloidosis, Hereditary, Transthyretin-Related

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study aims to determine the positive predictive value of incidental cardiac uptake on bone scintigraphy for diagnosing transthyretin cardiac amyloidosis, in patients who underwent scintigraphy for reasons other than suspected amyloidosis. The study is an observational, descriptive, multicenter, national study using retrospective data from routine care. Patients with incidental cardiac uptake will be recalled for further diagnostic assessment.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥ 18 years)
* Patients who underwent bone scintigraphy with 99mTc-HMDP/DPD/PYP for any indication
* Incidental cardiac uptake (Perugini grade ≥2) confirmed by a nuclear medicine specialist

Exclusion Criteria:

* Patients under legal protection
* Patients refusing the reuse of their data after individual information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent scintigraphy for reasons other than suspected amyloidosis
Sampling Method: Non-Probability Sample
Enrollment: 57 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Cardiac amyloidosis diagnosis | After the reassessment evaluation (one-day evaluation)

IPD SHARING:
Plan to Share IPD: No